CLINICAL TRIAL: NCT05554744
Title: Endoscopic Ultrasound-guided Fine-needle Injection for Multiple Endocrine Neoplasia Type 1-related Pancreatic Neuroendocrine Tumors: a Prospective Multicenter Study
Brief Title: EUS-FNI for MEN1-related Pancreatic Neuroendocrine Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Shanyu Qin, Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-K034-01
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Multiple Endocrine Neoplasia Type 1; Pancreatic Neuroendocrine Tumor
Keywords: Multiple endocrine neoplasia type 1; Pancreatic neuroendocrine tumor; Endoscopic ultrasonography-guided fine-needle injection; Ablation
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Adenoma, Islet Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEN1-1-related pNETs (Experimental): The patients with MEN1-1-related pNETs will undergo EUS-FNI with ethanol or lauromacrogol
  Interventions: Procedure: EUS-guided fine-needle injection

INTERVENTIONS:
Procedure: EUS-guided fine-needle injection — Diagnostic evaluation for suspected MEN1-1-related pNETs is conducted by cytology or immunohistochemistry and genetic testing. EUS-FNA is performed to obtain samples. After puncturing with the needle, ethanol/ lauromacrogol under the guidance of EUS was injected into the tumor The volume of ethanol/ lauromacrogol is administrated based on the tumor size.

SUMMARY:
The present study aims to evaluate the feasibility, safety and efficacy of EUS-FNI for MEN1-related pNETs

DETAILED DESCRIPTION:
The management of multiple endocrine neoplasia type 1 (MEN1-1)-related pancreatic neuroendocrine tumors (pNETs) remains controversial. In general, surgical resection is currently the first-line therapy for MEN1-1-related pNETs. However, the surgical resection of pNETs is conditional for specific patients, and the incidence of postoperative adverse events is still high. Recently, several studies have demonstrated that endoscopic ultrasonography (EUS)-guided fine-needle injection (EUS-FNI) with ethanol or lauromacrogol may provide an alternative to surgical resection of pNETs. Nevertheless, their sample size was relatively small and conclusions were drawn based on short-term results. Therefore, a multicenter prospective study is being performed to further access the efficacy and safety of EUS-FNI for MEN1-1-related pNETs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MEN1-1-related pNETs are evaluated by histopathology and genetic testing.
2. Patients who refuse surgery.
3. Patients who have given their fully informed consent.

Exclusion Criteria:

1. Patients who are not suitable for the endoscopic procedure.
2. Patients who have blood coagulation dysfunction, mental disorders, mild or severe cardiorespiratory.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of blood glucose level | Within 7 days of the last ablation and every 6 months up to 24 months
  Changes in the lowest blood glucose levels between baseline and last treatment and each study visit
Changes of insulin level | Within 7 days of the last ablation and every 6 months up to 24 months
  hanges in the insulin levels between baseline and last treatment and each study visit
Changes of C peptide | Within 7 days of the last ablation and every 6 months up to 24 months
  Changes in the C peptide levels between baseline and last treatment and each study visit
Imaging response | Every 6 months up to 24 months
  Complete ablation on the CE-CT or CE-EUS

SECONDARY OUTCOMES:
Feasibility of EUS-FNI | At the time of procedure
  The success rate of EUS-FNI
Safety of EUS-FNI | Within 1 month after treatment
  The occurrence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shanyu Qin, Ph.D, Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Yes